CLINICAL TRIAL: NCT05856695
Title: A Phase II Study Assessing the Efficacy of Etoposide Free Chemotherapy Plus Durvalumab (MEDI4736) in First Line Extensive Disease Small Cell Lung Cancer (SCLC)
Brief Title: Durvalumab Plus Etoposide-free Chemotherapy in First-line Treatment of Extensive-disease Small-sell Lung Cancer (SCLC)
Acronym: TAXIO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-2203
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: IFCT; SCLC; SCLC Extensive Stage
MeSH Terms: interventions — Carboplatin; Paclitaxel; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carboplatin + Paclitaxel + Durvalumab (Experimental): Carboplatin AUC 6, day 1 of three-week cycle for four cycles Paclitaxel 200 mg/m² day 1 of a three-week cycle for four cycles Durvalumab 1500 mg every 3 weeks for 4 cycles followed by 1500 mg maintenance every 4 weeks until progression, unacceptable toxicity, or consent withdrawal
  Interventions: Drug: Carboplatin + Paclitaxel + Durvalumab

INTERVENTIONS:
Drug: Carboplatin + Paclitaxel + Durvalumab — Carboplatin AUC 6, day 1 of three-week cycle for four cycles Paclitaxel 200 mg/m² day 1 of a three-week cycle for four cycles Durvalumab 1500 mg every 3 weeks for 4 cycles followed by 1500 mg maintenance every 4 weeks until progression, unacceptable toxicity, or consent withdrawal

SUMMARY:
The current study is intended to be a "proof of concept" to evaluate the potential value of synergy between paclitaxel carboplatin and immunotherapy. If a signal clearly shows superiority over the CASPIAN data , we will have arguments to think that the combination of paclitaxel and carboplatin is more suitable for synergy with immunotherapy than the standard etoposide and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent.

   * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
   * Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
2. Patients diagnosed with histologically confirmed SCLC
3. Extended-Stage Disease at time of accrual according to the criteria of the Veteran's Administration Lung Cancer Group (VALG). Extended disease is defined as going beyond hemithorax and supraclavicular ganglionic areas, and malignant pleural effusions will be considered extended diseases.
4. At least one measurable target lesion according to RECIST v1.1 per investigator assessment.The radiological assessment has to be done within the timelines indicated.
5. Age ≥ 18 years.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 (see Appendix 1).
7. Body weight >30 kg.
8. Adequate biological functions:

   * Creatinine clearance ≥ 45 ml/min (Cockroft or MDRD or CKD-epi);
   * Hemoglobin ≥ 9.0 g / dL
   * Neutrophils ≥ 1500 /μL
   * Platelets ≥ 100 000 /μL
   * Bilirubin ≤ 1.5 x normal except for patients with proved Gilbert syndrome (≤ 3 x ULN)
   * ALT and AST ≤ 2.5 x normal upper value except in case of liver metastases (≤ 5 x normal upper value).
9. Woman patients who are no longer likely to procreate (physiologically unfit to carry a pregnancy), which includes:

   * Hysterectomy
   * Ovariectomy
   * Bilateral tubal ligation
   * Postmenopausal women:

     * Patients not using hormone replacement therapy should have had a complete cessation of menstruation for at least one year and be over 45 years old, or, if in doubt, have an FSH (Follicle Stimulating Hormone)> 40 mIU/mL and a Estradiol value<40 μg/mL (<150 pmol/L)
     * Patients using hormone replacement therapy should have had a complete cessation of menstruation for at least one year and be over 45 years of age or have evidence of menopause (FSH and estradiol levels) prior to initiation of hormone replacement therapy.

   Woman patients who are of childbearing potential are eligible:
   * They must have a negative serum pregnancy test within the week preceding the first dose of treatment and preferably as close as possible to the first dose.
   * They must agree to use methods of contraception acceptable for IFCT, when used in accordance with the product leaflet and the doctor's instructions, are as follows:

     * An intrauterine device with a failure rate of less than 1% per year
     * Male sterilized partner (vasectomy with azoosperm documentation) prior to inclusion of the patient and who is the sole partner of the patient.
     * Total abstinence from sexual intercourse 14 days before the start of treatment, throughout the duration of treatment and at least 21 days after the last dose of treatment.
     * Double-barrier contraception: condom and cape (diaphragm or cervical / vaginal cap) with a vaginal spermicidal agent (foam / gel / film / cream / suppository).
     * Oral, combined or progestin contraceptive alone.
     * Injectable progestin.
     * Levonorgestrel implant.
     * Vaginal ring impregnated with estrogen.
     * Percutaneous contraceptive patch. Contraceptive methods should be used throughout the course of treatment and should be maintained for 6 months after the end of treatment.
10. Male subjects who are sexually active with a woman of childbearing potential are eligible if an efficacious contraception method should be used during the treatment and during the 6 months following the last dose.
11. Patient must have a life expectancy of at least 12 weeks.
12. Patient covered by a national health insurance.

Exclusion Criteria:

1. Non-small cell lung cancer (NSCLC) or combined SCLC and NSCLC.
2. Prior systemic anticancer therapy for SCLC.
3. Radiotherapy needed at initiation of treatment.
4. Major surgical procedure (as defined by the Investigator) within 28 days prior initiation of treatment.

   Note: Local surgery of isolated lesions for palliative intent is acceptable.
5. Symptomatic brain metastasis. Note: patient with asymptomatic or treated and stable brain metastasis for at least 1 month prior to study treatment are eligible. Patients with suspected brain metastases at screening should have a CT/MRI of the brain prior to study entry.
6. History of leptomeningeal carcinomatosis.
7. Symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, cardiac arrhythmia or clinically uncontrolled heart disease.
8. Mean QT interval corrected (QTc) ≥470 ms.
9. Corticosteroid therapy at a dose greater than 10 mg per day of prednisolone or equivalent for more than 10 days within 14 days prior initiation of treatment.

   Note: Intranasal, inhaled, topical steroids, or local steroid injections and steroids as premedication for hypersensitivity reactions are allowed.
10. Serum sodium <125 mmol/L unless corrective treatment prior to initiation of study treatment.
11. Hypercalcemia despite corrective treatment (corrected calcemia = Calcium (mmol) + [(40- albumin (g)) x 0.025]).
12. History of allogenic organ transplantation.
13. Immunosuppressive systemic therapy (cyclophosphamide, aziathioprine, methotrexate, thalidomide and TNF inhibitor) within 28 days prior to inclusion.
14. Active or prior documented autoimmune disease or inflammatory disorders including but is not limited to inflammatory bowel disease (colitis or Crohn's disease), diverticulitis (with the exception of diverticulosis), sarcoidosis syndrome, myasthenia gravis, lupus erythematosus, rheumatoid arthritis, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain Barré's syndrome, multiple sclerosis, vasculitis and glomerulonephritis. Patients with severe psoriasis (10% of your body's surface area) are not eligible.

    Note: The following are exceptions are listed below:
    * patients with vitiligo or alopecia,
    * patients with history of autoimmune hypothyroidism treated with a stable dose of hormone replacement therapy,
    * any chronic skin condition that does not require systemic therapy,
    * patients without active disease in the last 5 years may be included but only after consultation with the investigator,
    * patients with celiac disease controlled by diet alone,
    * patients with diabetes treated with insulin.
15. Serious chronic gastrointestinal conditions associated with diarrhea
16. History of idiopathic pulmonary fibrosis, organized pneumonia (i.e., bronchiolitis obliterans), drug-induced pulmonary pathology or active signs of pneumonia, interstitial lung disease (whatever the cause) detected on the pulmonary CT-scan.
17. History of cancer Note: Patients with a history of cancer for more than 3 years are eligible if they have been treated and considered cured. Patients with a history of basal cell carcinoma of the skin or in situ carcinoma of the cervix are eligible.
18. Concomitant anti-cancer treatment or within 3 years prior to the start of study treatment, including chemotherapy, immunotherapy, hormone therapy, biotherapy or anti-angiogenic treatment (VEGF inhibitors or VEGFR inhibitors).
19. Any medical or personal that would make the patient unable to comply with study procedures and/or could interfere with the patient safety.
20. Receipt of live, attenuated vaccine within 30 days prior to the first dose of study drugs.

    Note: Patients, if enrolled, should not receive live vaccine whilst receiving study drugs and up to 30 days after the last dose of study drugs. Nucleic acid vaccines, inactivated vaccines against COVID-19 are allowed.
21. Ongoing or active infection including:

    * COVID-19.
    * Tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice).
    * Hepatitis B virus (known positive HBV surface antigen [HbsAg] result). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible.
    * Positive hepatitis C virus (HCV).
22. Patients with a known history of a positive test for HIV or known AIDS who have not received effective antiretroviral therapy (ART) for the last 4 weeks and who have an HIV viral load >200 copies/mL, regardless of CD4+ T-cell count. Paraneoplastic syndrome (PNS) of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents) or clinical symptomatology suggesting worsening of PNS.
23. Pregnant or lactating woman. Note: Women who are breastfeeding should stop breastfeeding before the first dose of treatment, throughout the course of treatment and at least 3 months after the last dose of treatment.
24. Known allergy or hypersensitivity to study treatment or any excipient.
25. Concomitant treatment with another experimental treatment or participation in another clinical trial.
26. Patient who is subject to legal protection or who is unable to express his will.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | At 12 months
  Overall Survival (OS) defined as the time from the date of first dose of study drug to the date of death due to any cause

SECONDARY OUTCOMES:
Best response rate (RECIST 1.1) | About 48 months
  Best response rate (RECIST 1.1) which is defined as the percentage of subjects with a complete response (CR) or partial response (PR) determined by Investigator review and by independent reviewer as per RECIST v1.1 criteria.
Overall Survival (OS) | About 48 months
  Overall Survival (OS) defined as the time from the date of first dose of study drug to the date of death due to any cause
Overall Survival (OS) | At 24 months
  Overall Survival (OS) defined as the time from the date of first dose of study drug to the date of death due to any cause
Overall Survival (OS) | At 36 months
  Overall Survival (OS) defined as the time from the date of first dose of study drug to the date of death due to any cause
Progression free survival (PFS) | About 48 months
  Progression free survival (PFS) defined as the time from the date of inclusion to the earliest date of disease progression, as determined by Investigator review and by independent reviewer of radiographic disease assessments per RECIST v1.1, or death due to any cause
Safety and tolerability of paclitaxel carboplatin and durvalumab. | About 48 months
  Incidence, nature, and severity of adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Quality of life of patients | About 48 months
  Change from baseline of Quality of life assessment using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30 LC13) at all scheduled time points.

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - Abbeville - CH, Abbeville
  - Amiens - Clinique de l'Europe, Amiens
  - Angers - CHU, Angers
  - Besançon - CHU, Besançon
  - Bordeaux - CHU, Bordeaux
  - Boulogne - Ambroise Paré, Boulogne-Billancourt
  - Caen - CHU Côte de Nacre, Caen
  - Chambéry - CH, Chambéry
  - Cholet - CH, Cholet
  - Colmar - CH, Colmar
  - Annemasse - CH, Contamine-sur-Arve
  - Créteil - CHI, Créteil
  - Dijon - CHU Bocage, Dijon
  - Grenoble - CHU, Grenoble
  - Le Mans - CHG, Le Mans
  - Lyon - URCOT, Lyon
  - Marseille - APHM, Marseille
  - Marseille - Hôpital Européen, Marseille
  - CHU Montpellier, Montpellier
  - Morlaix - CH, Morlaix
  - Orléans - CHR, Orléans
  - Paris - Bichat, Paris
  - Paris - Hôpital Cochin, Paris
  - Paris - Tenon, Paris
  - Rennes - CHU, Rennes
  - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Toulon - Sainte Anne HIA, Toulon
  - CHU Toulouse, Toulouse
  - Tours - CHU, Tours
  - Vandoeuvre-lès-Nancy - CRLCC, Vandœuvre-lès-Nancy
  - Villefranche sur Saône - CH, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Undecided